CLINICAL TRIAL: NCT05744076
Title: Analysis of Circulating Exosomes in Melanoma Patients
Acronym: EXOMEL1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/401
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis is that PD-L1[Programmed Death-Ligand 1] labeling in exosomes could be a biomarker of disease progression in melanoma. The rate of circulating exosomes, their size and the exosomal expression of PD-L1 could be correlated with the stage of the disease, the response to treatment and/or the prognosis of patients. In this study, blood samples (EDTA tubes taken as part of routine care at Besançon University Hospital) and associated clinical data are reused.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma patients admitted in Besançon University Hospital
* exigible for immunotherapy such as anti PD-L1/PD-1
* Age ≥18 years
* Affiliation to a social security system,

Exclusion Criteria:

* Minor patients
* Patients who have expressed their opposition to the reuse of their data and biological samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Melanoma patients admitted in Besançon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of circulating exosomes | Day 1
  Dosage of proteic biomarkers in circulating exosomes, plasma and tumor tissues. Blood samples were taken in standard care, before initiation of immunotherapy and then during disease follow-up until progression and tumor evaluation

SECONDARY OUTCOMES:
PDL1 marking | Day 1
  Compare PD-L1 labeling in exosomes to PD-L1 labeling in plasma and in tumor tissue. Blood samples were taken in standard care, before initiation of immunotherapy and then during disease follow-up until progression and tumor evaluation
Other proteins detection | Day 1
  Identify other proteins of interest in circulating exosomes. Blood samples were taken in standard care, before initiation of immunotherapy and then during disease follow-up until progression and tumor evaluation.
Determine whether the initial exosome concentration (at T0) is associated with a response to treatment. | Day 1
  Dosage of PD-L1 in circulating exosomes. Blood samples were taken in standard care, before initiation of immunotherapy and then during disease follow-up until progression and tumor evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

REFERENCES:
- [Derived] Nardin C, Vautrot V, Naiken I, Doussot A, Puzenat E, De Girval C, Garrido C, Aubin F, Gobbo J. Monitoring Pseudoprogression Using Circulating Small Extracellular Vesicles Expressing PD-L1 in a Melanoma Patient Treated With Immune Checkpoint Inhibitors. J Extracell Biol. 2025 Jun 22;4(6):e70066. doi: 10.1002/jex2.70066. eCollection 2025 Jun. PMID 40552104